CLINICAL TRIAL: NCT06081829
Title: A Phase 2, Open-label, Multicenter Study of Orally Administered Ivosidenib in Previously Treated Japanese Subjects With Nonresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Brief Title: A Phase 2 Study of Ivosidenib in Previously Treated Japanese Subjects With Nonresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95031-008
Record Dates: First submitted 2023-09-14; First posted 2023-10-13 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Cholangiocarcinoma Non-resectable; Cholangiocarcinoma Metastatic
Keywords: IDH-1 Mutation; Cholangiocarcinoma Non-resectable with an IDH-1 Mutation; Cholangiocarcinoma Metastatic with an IDH-1 Mutation
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label Ivosidenib (Experimental): 250 mg Tablets
  Interventions: Drug: Ivosidenib

INTERVENTIONS:
Drug: Ivosidenib — Subjects will take 2 tablets (500 mg total) orally once daily.

SUMMARY:
This study will enroll participants with nonresectable or metastatic cholangiocarcinoma with an Isocitrate dehydrogenase protein, 1 (IDH1) mutation, who have previously received at least 1, but no more than 2, prior regimens for advanced disease. All participants will receive ivosidenib daily throughout multiple 28 day cycles. Study treatment will be administered until participant experiences unacceptable toxicity, disease progression, or other discontinuation criteria are met. Study visits will be conducted every week during Cycle 1 (Days 1, 8, 15, and 22), every other week during Cycles 2 and 3, and Day 1 of each cycle thereafter. After the last dose of treatment, participants will attend an end of treatment and a post-treatment follow-up visit, and participants will be followed to assess overall survival. Study visits may include a tumor assessment, physical exam, electrocardiogram (ECG), blood and urine analysis, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Have nonresectable or metastatic cholangiocarcinoma and are not eligible for curative resection, transplantation or ablative therapies
* Have documented IDH1 gene-mutated disease from a tumor biopsy
* Have an ECOG PS score of 0 or 1
* Have an expected survival of 3 months or more
* Have at least one evaluable and measurable lesion
* Have disease progression following the most recent of 1 or 2 prior systemic regimens for advanced disease with progression on the treatment that was most recently given at a minimum, and must have received at least 1 gemcitabine- or 5-FU -containing regimen
* Have recovered from side effects associated with the prior treatment therapy
* Have adequate bone marrow function
* Have adequate hepatic (liver) and renal (kidney) function
* Women of child bearing potential must have a negative serum pregnancy test before starting study treatment, and use birth control during the study and for 90 days after the last dose of ivosidenib
* Fertile men with female partners of child bearing potential must use birth control during the study and for 90 days after the last dose of ivosidenib

Exclusion Criteria:

* Received a prior IDH inhibitor.
* Have known symptomatic brain metastases requiring steroids.
* Pregnancy, possibility of becoming pregnant during the study and breast-feeding women or woman who plans to restart breast-feeding after the study drug administration/intake.
* Are taking known strong cytochrome P450 (CYP) 3A4 inducers or sensitive CYP3A4 substrate medications with a narrow therapeutic window
* Have significant heart disease, including congestive heart failure, myocardial infarction (heart attack) unstable angina (chest pain) and/or stroke, within 6 months before starting the study
* Have a heart-rate corrected QT interval ≥450 msec or other factors that increase the risk of QT prolongation or arrhythmic events
* . Have active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis (paralysis of the stomach), or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Have known medical history of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - National Cancer Center Hospital East (JPN-002), Kashiwa
  - Kumamoto University Hospital (JPN-004), Kumamoto
  - National Hospital Organization Shikoku Cancer Center (JPN-007), Matsuyama
  - Osaka International Cancer Institute (JPN-005), Osaka
  - Hokkaido University Hospital (JPN-006), Sapporo
  - National Cancer Center Hospital (JPN-001), Tokyo
  - Kanagawa Cancer Center (JPN-003), Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label Ivosidenib
Started | 12
Completed | 0 (Study is still ongoing, and participants are still on-study as noted under the "Reason Not Completed" section.)
Not Completed | 12
Not completed — Participants still on-study | 8
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Age, Continuous [Median (Standard Deviation); unit: years] | 61.5 (12.27)
Age, Customized [Count of Participants; unit: Participants]
  45-<65 years old | 7
  >=65 years old | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression Free Survival (PFS) Rate
Description: Proportion of subjects who are alive and progression-free (using RECIST v1.1) at 6 months after Day 1 (C1D1) per Independent Radiology Center (IRC)
Time Frame: Through 6 months after the first dose
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
percentage of participants | 25.0 [8.1 to 46.5]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from Day 1 to the date of first documentation of disease progression as assessed by the Investigator and by the IRC per RECIST v1.1. or death due to any cause
Time Frame: Approximately 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
months | 4.21 [2.69 to NA] — Data was not estimable (survival time exceeds the longest observed or censored survival time as of the data cut-off date)

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Approximately 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
months | NA [5.19 to NA] — Data was not estimable (median survival time exceeds the longest observed or censored survival time as of the data cut-off date)

4. Secondary Outcome: Objective Response (OR) Rate
Description: Complete response or partial response
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: The time from date of first documented confirmed complete response (CR) or confirmed partial response (PR) to date of first documented disease progression or death due to any cause
Time Frame: Approximately 1 year
Population: No participants achieved a complete response or partial response, and therefore there were no participants who could be assessed for their duration of response.
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Response (TTR)
Description: The time from Day 1 to date of first documented confirmed complete response (CR) or confirmed partial response (PR)
Time Frame: Approximately 1 year
Population: No participants achieved a complete response or partial response, and therefore there were no participants who could be assessed for their time to response.
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Health-Related Quality of Life Using EORTC-QLQ-C30 Questionnaire Scores.
Description: The European Organisation for Research and Treatment of Cancer - Quality Of Life Questionnaire - Core Questionnaire (EORTC-QLQ-C30) is comprised of 5 functional scales ((Physical functioning, Role functioning, Cognitive functioning, Emotional functioning and Social functioning), 3 symptom scales (Fatigue, Pain and Nausea/Vomiting), 6 additional single items (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties) and global health status (GHS). All of the scale scores range from 0 - 100; for the functional scales and GHS the higher score represents better functioning and for the symptom scales and single items the higher score represents an increase in symptoms.
  .
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 9
score on a scale
  Physical Functioning | -6.7 (15.63)
  Role Functioning | -9.3 (16.90)
  Cognitive Functioning | -1.9 (10.02)
  Emotional Functioning | -8.3 (18.63)
  Social Functioning | -14.8 (17.57)
  Fatigue | 7.4 (16.67)
  Pain | 7.4 (32.39)
  Nausea/Vomiting | 7.4 (12.11)
  Dyspnea | 22.2 (40.82)
  Insomnia | 18.5 (29.40)
  Appetite Loss | 7.4 (32.39)
  Constipation | -7.4 (14.70)
  Diarrhea | 3.7 (20.03)
  Financial Difficulties | 0.0 (23.57)
  GHS | -20.4 (22.48)

8. Secondary Outcome: Change From Baseline in Health-Related Quality of Life Using EORTC-QLQ-BIL21 Questionnaire Scores.
Description: The European Organisation for Research and Treatment of Cancer - Quality Of Life Questionnaire - Cholangiocarcinoma and Gallbladder Cancer Module (EORTC-QLQ-BIL21) scores range from 0 - 100 with higher scores representing more severe symptoms.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 9
score on a scale | 8.3 (12.50)

9. Secondary Outcome: Average EQ-5D-5L VAS Scores
Description: The 5-level EuroQol five dimensions questionnaire (EQ-5D-5L) visual analogue scale (VAS) scores range from 0 to 100 with a higher number representing a better health status.
Time Frame: Baseline, Cycle 3 Day 1 (cycle = 28 days), and End of Treatment Visit (within 5 to 33 days after last dose of treatment, approximately 1 year total)
Population: The number analyzed differs due to missing participant data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
score on a scale
  Baseline | 78.8 (10.80)
  Cycle 3 Day 1: number analyzed (Participants) | 11
  Cycle 3 Day 1 | 75.8 (15.61)
  End of Treatment: number analyzed (Participants) | 9
  End of Treatment | 61.7 (27.05)

10. Secondary Outcome: Total Number of Adverse Events (AEs)
Time Frame: Approximately 1 year
Measure: Number; unit: Number of Adverse Events
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Number of Adverse Events | 24

11. Secondary Outcome: Total Number of Participants With Adverse Events (AEs) Leading to Dose Modifications
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants | 0

12. Secondary Outcome: Total Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants | 0

13. Secondary Outcome: Total Number of Participants With Serious Adverse Events (SAEs)
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants | 2

14. Secondary Outcome: Total Number of Participants With Adverse Events (AEs) Leading to Death
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants | 0

15. Secondary Outcome: Average Area Under the Concentration-vs Time Curve From 0 to Time of Last Measurable Concentration (AUC0-t)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1
Population: One participant was excluded from Cycle 2 Day 1 data analysis since their dose was reduced.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
ng*h/mL
  Cycle 1 Day 1 | 18699 (43.5)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 22404 (27.4)

16. Secondary Outcome: Average AUC Over 1 Dosing Interval at Steady State (AUCtau,ss)
Time Frame: Cycle 2 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 11
ng*h/mL | 74121 (30.0)

17. Secondary Outcome: Average Time to Maximum Concentration (Tmax)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1
Population: One participant's data was excluded from Cycle 2 Day 1 since the ivosidenib dose was reduced.
Measure: Median (Full Range); unit: hours
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
hours
  Cycle 1 Day 1 | 2.98 [1.85 to 5.93]
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 3.83 [1.83 to 3.97]

18. Secondary Outcome: Average Maximum Concentration (Cmax)
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1
Population: One participant's data was excluded from Cycle 2 Day 1 since the ivosidenib dose was reduced.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
ng/mL
  Cycle 1 Day 1 | 4918 (42.7)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 4781 (22.8)

19. Secondary Outcome: Average Trough Concentration (Ctrough)
Time Frame: Cycle 2 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 11
ng/mL | 2058 (28.7)

20. Secondary Outcome: Average Plasma 2-hydroxyglutarate (2-HG) Concentrations
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1
Population: One participant's data was excluded from Cycle 2 Day 1 since the ivosidenib dose was reduced.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
ng/mL
  Cycle 1 Day 1 | 597 (532.07)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 79.95 (41.166)

21. Secondary Outcome: Number of Participants With no Change, Plus 1 or Plus 2 Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status (ECOG PS) Score
Description: From baseline to worst value of post-baseline assessments. ECOG PS scores range from 0 to 5 with 0 representing a person being fully active and 5 being the patient is dead.
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ivosidenib
Number analyzed (Participants) | 12
Participants
  Baseline Score of 0 and Worst Post-Baseline Score of 0 (no change) | 7
  Baseline Score of 0 and Worst Post-Baseline Score of 1 (+1 change) | 2
  Baseline Score of 0 and Worst Post-Baseline Score of 2 (+2 change) | 1
  Baseline Score of 1 and Worst Post-Baseline Score of 1 (no change) | 2

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Description: Adverse events will be assessed during study visits.
Arm/Group | Open-Label Ivosidenib
All-Cause Mortality (participants affected / at risk) | 4/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Ivosidenib (N=12)
Electrocardiogram QT prolonged (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Ivosidenib (N=12)
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT06081829/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT06081829/SAP_001.pdf